CLINICAL TRIAL: NCT04410653
Title: Afatinib in Advanced NRG1-Rearranged Malignancies: the NCT/DKTK PMO-1604 Phase-II Trial
Brief Title: Afatinib in Advanced NRG1-Rearranged Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: German Consortium for Translational Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT/DKTK PMO-1604
Record Dates: First submitted 2020-05-15; First posted 2020-06-01 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Metastatic and Locally Advanced NRG1-rearranged Malignancies
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (KRASwt PDAC) (Experimental)
  Interventions: Drug: Afatinib 40 MG
- Arm 2 (IMA) (Experimental)
  Interventions: Drug: Afatinib 40 MG
- Arm 3 (other) (Experimental)
  Interventions: Drug: Afatinib 40 MG

INTERVENTIONS:
Drug: Afatinib 40 MG — single oral dose of afatinib each day starting at a dose of 40 mg on day 1, continuously, until the development of progressive disease or unacceptable adverse events

SUMMARY:
Whole-genome and transcriptome sequencing of patients with advanced solid tumors enrolled in the NCT/DKTK MASTER (Molecularly Aided Stratification for Tumor Eradication Research) program revealed recurrent NRG1 fusions in a substantial proportion of patients with KRAS wild-type (KRASwt) pancreatic adenocarcinoma (PDAC) and a case of signet-ring cell carcinoma of the appendix. NRG1 rearrangements drive tumor development through ERBB receptor-mediated signaling, as evidenced by objective response to ERBB inhibition in two cases of NRG1-rearranged PDAC in the MASTER cohort. Recently, NRG1 fusions have also been identified as a therapeutic target in a substantial number of the invasive mucinous subtype of lung adenocarcinoma (IMA) as well as in cholangiocellular carcinoma and, at low incidence, other tumor entities, suggesting oncogenic properties across a broader spectrum of malignancies.

Within this phase II clinical trial, the investigators aim to investigate the efficacy of the pan-ERBB inhibitor afatinib in advanced-stage NRG1-rearranged malignancies across all tumor entities following progression on standard therapy. Due to the enrichment of NRG1-rearrangements observed in KRASwt PDAC and IMA, two separate study arms will focus on these tumor entities while a third arm will allow inclusion of patients with any other NRG1 rearranged malignancy. Recruitment of adequate patient numbers in this well-defined molecular subgroup will be achieved by a multicenter approach including all DKTK partner sites and on-site pre-screening of PDAC for KRAS mutational status. Eligible patients will be identified by in-depth molecular characterization of tumors within the NCT/DKTK MASTER program or identification of a NRG1-rearranged tumor by another method for fusion detection (e.g. gene fusion panel).

Patients with NRG1-rearranged tumors fulfilling eligibility criteria will be offered to participate in the trial and receive afatinib monotherapy until tumor progression or discontinuation for other reasons. To assess mechanisms of secondary resistance and to investigate the clinical impact of liquid biopsies in this setting, blood samples for exome sequencing will be taken prior to initiation of the study treatment as well as at the time of progression.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a written informed consent
2. Patient is able to understand and comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
3. Progressive metastatic or locally advanced NRG1-Rearranged Malignancy as determined by investigator
4. At least one measurable lesion that can be accurately assessed at baseline by CT or MRI and is suitable for repeated assessment
5. Prior administration of at least one standard treatment for primary and/or relapsed malignancy according to current guidelines
6. Eastern Cooperative Oncology Group Performance Status ≤ 1
7. Male or female patient aged ≥ 18, no upper age limit
8. Postmenopausal or evidence of non-childbearing status. For women of childbearing potential: negative urine pregnancy test at baseline and highly effective forms of contraception in place thereafter as well as confirmed negative urine pregnancy test prior to treatment on day 1 of every cycle and at end of treatment period.

   Evidence of childbearing potential is defined as:

   o Fertile, following menarche and until becoming post-menopausal unless permanently sterile

   Postmenopausal or evidence of non-childbearing status is defined as:
   1. Amenorrheic for 1 year or more without an alternative medical cause following cessation of exogenous hormonal treatments PLUS Follicle stimulating hormone (FSH) levels in the postmenopausal range in women not using hormonal contraception or hormonal replacement therapy
   2. Surgical sterilisation (bilateral oophorectomy, hysterectomy or bilateral salpingectomy)
9. Female patients of child bearing potential and male patients with partners of child bearing potential, who are sexually active, must agree to the use of two highly effective forms of contraception. This should be started from the signing of the informed consent and continue throughout period of taking study treatment and for 1 month (female patients) / 3 months (male patients) after last dose of study drug.
10. Identification of NRG1 rearrangements within NCT/DKTK MASTER (Heidelberg Ethics Committee Reference No.: S-206/2011) or identification of a NRG1 fusion by another method for fusion detection (e.g. gene fusion panel)
11. Adequate bone marrow, renal, and hepatic function defined by laboratory tests within 14 days prior to study treatment:

    1. Absolute neutrophil count (ANC) ≥1500 / mm3. (ANC >1000/mm3 may be considered in special circumstances such as benign cyclical neutropenia as judged by the investigator and in discussion with the sponsor).
    2. Platelet count ≥75,000 / mm3.
    3. Estimated creatinine clearance > 45ml / min (according to Crockroft-Gault-formula).
    4. Total Bilirubin ≤ 1.5 times upper limit of normal (Patients with Gilbert's syndrome total bilirubin must be ≤4 times institutional upper limit of normal (ULN)).
    5. Aspartate amino transferase (AST) or alanine amino transferase (ALT) ≤ three times the ULN (if related to liver metastases ≤ five times ULN).
12. Left ventricular function with resting ejection fraction ≥ 50% or above the LLN.
13. Recovered from any previous therapy related toxicity to ≤Grade 1 at study entry (except for stable sensory neuropathy ≤Grade 2 and alopecia)
14. Written informed consent that is consistent with ICH-GCP guidelines

Exclusion Criteria:

1. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years
2. Concurrent or previous treatment within 4 weeks in another interventional clinical trial with an investigational anticancer therapy
3. Prior treatment with afatinib
4. Hormonal treatment within 2 weeks prior to start of study treatment (continued use of anti-androgens and/or gonadorelin analogues for treatment of prostate cancer permitted)
5. Radiotherapy within 4 weeks prior to randomization , except as follows:

   i.) Palliative radiation to target organs may be allowed up to 2 weeks prior to randomisation, and

   ii.) Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with coordinating investigator/ scientific investigator prior to enrolling.
6. Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
7. Known hypersensitivity to afatinib or the excipients of any of the trial drugs
8. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of ≥ 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to randomisation.
9. Women of child-bearing potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly prior to study entry, for the duration of study participation and for 1 month (female patients)/ 3 months (male patients) after last dose of study drug (after EOT).
10. Women who are pregnant, nursing, or who plan to become pregnant while in the trial
11. Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug
12. Known pre-existing interstitial lung disease (ILD)
13. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhoea, malabsorption)
14. Leptomeningeal carcinomatosis
15. Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids, anti-convulsants or have been on stable dose of corticosteroids for at least 4 weeks before starting study treatment. Any symptoms attributed to brain metastases must be stable for at least 4 weeks before starting study treatment.
16. Persistent toxicity (≥Grade 2 according to Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) caused by previous cancer therapy, excluding alopecia
17. Clinical signs of active infection (>Grade 2 according to CTCAE version 5.0)
18. History of HIV infection and immunocompromised patients
19. Viral active or chronic hepatitis (HBV or HCV)
20. Dementia or significant impairment of cognitive state
21. Epilepsy requiring pharmacologic treatment
22. Heart failure NYHA III/IV
23. Severe obstructive or restrictive ventilation disorder
24. Concomitant use of P-gp- inhibitors (e.g. ritonavir, ciclosporin A, ketoconazole, itraconazole, erythromycin, verapamil, quinidine, tacrolimus, nelfinavir, saquinavir, amiodarone) and BCRP inhibitors (e.g. rosuvastatin, sulfasalazine). The required washout period prior to starting afatinib is at least five half-lifes.
25. Concomitant use of P-gp-inducers (e.g. rifampicin, carbamazepine, phenytoin, phenobarbital, St. John's wort) The required washout period prior to starting afatinib is at least five half-lifes (e.g. 5 weeks for phenobarbital).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate | 6 months
  Primary objective of the study is to assess clinical activity of afatinib in adult patients with (locally) advanced or recurrent solid tumors harboring NRG1-rearrangments. Clinical efficacy is determined by disease control rate (DCR) including CR, PR, and SD according to RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Progression-free Survival | through study completion, an average of 1 year
  To assess progression-free survival (PFS) of afatinib in adult patients with advanced solid tumors harboring NRG1-rearrangments.
Overall survival | through study completion, an average of 1 year
  To assess OS (overall survival) of afatinib in adult patients with advanced solid tumors harboring NRG1-rearrangments.
Safety and Tolerability: Toxic effects are graded according to the National Cancer Institute Common Toxicity Criteria (CTCAE) version 5.0 | 6 months
  This endpoint includes all AEs, their severity, SAEs, the relation of AEs to the study treatment, dose modifications for toxicity and discontinuation of study treatment during the trial phase. Toxic effects are graded according to the National Cancer Institute Common Toxicity Criteria (CTCAE) version 5.0.
Patient reported Outcomes | 6 months
  Patient Reported Outcomes including quality of life (QLQ) of patients treated with afatinib.
  Patient-Reported Outcomes (PROs) including health-related quality of life (QoL) are calculated as the new European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 Summary Score recommended by the EORTC Quality of Life Group. In addition, the EORTC QLQ function and symptom scores will be calculated according to the actual EORTC Scoring Manual.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Heining, Dr., Principal Investigator — National Center of Tumor Diseases (NCT) Dresden
Locations (2):
- Germany (2):
  - NCT Dresden, Dresden
  - NCT Heidelberg, Heidelberg

IPD SHARING:
Plan to Share IPD: Yes